CLINICAL TRIAL: NCT05639491
Title: The Petro-trigeminal Line: a Simple Radiological Marker for the Diagnosis of Cephaloceles of the Petrous Apex on MRI
Brief Title: Petro-trigeminal Line and Petrous Apex Cephaloceles
Acronym: APEX
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7960
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-11

CONDITIONS: Petrous Apex Meningioma
Keywords: Petrous apex cephaloceles; Petrous apex; meckel's cave; cavum-trigeminale-cephaloceles; arachnoïd kyst; meningoceles; trigeminal nerves
MeSH Terms: conditions — Meningocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
cephaloceles are rare lesions of the petrous apex, inconsistently listed as meningoceles or arachnoid cysts. They're consistent with a herniation posterolateral of the Meckel cavum within the petrous apex. These lesions may be the cause of a symptomatology varied, or be discovered by chance in subjects who have not been asymptomatic. Currently, there is no evidence in the literature a simple, fast and reproducible radiological marker that allows for the diagnosis of cephaloceles of the petrous apex, in particular the small ones. The purpose of this study is to validate a radiological benchmark simple and reproducible, the trigeminal petrol line, in order to improve the diagnosis of petrous apex cephaloceles

ELIGIBILITY:
Inclusion criteria:

* Major subjects (≥18 years old)
* patients who underwent an MRI with high resolution 3D T2 sequence between 01/01/2003 and 09/31/2020:
* 200 patients consulting for ENT pathology such as vertigo
* 9 patients presenting the radiological criteria in MRI of a cephalocele of the petrous apex according to the current data of the literature on a T2 3D HR sequence
* - Subject who has not expressed his opposition, after being informed, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Kinetic Artifacts
* Subject under guardianship or curatorship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subjects (≥18 years old) who underwent an MRI with high resolution 3D T2 sequence between 01/01/2003 and 09/31/2020:
  * consulting for ENT pathology such as vertigo
  * or presenting the radiological criteria in MRI of a cephalocele of the petrous
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Validate a radiological landmark allowing MRI diagnosis cephaloceles of the petrous apex | Files analysed retrospectively from from January 01, 2003 to September 31, 2020 will be examined
  This mark corresponds to the projection of a line drawn on an axial section, in the plane of the posterior roots of the trigeminal nerves, between the anterior and external edges of the petrous apex along the petro-trigeminal angle on each side.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie 1 - CHU de Strasbourg - France, Strasbourg, France